CLINICAL TRIAL: NCT06420882
Title: Comparison of Different Treatment Methods in Patella Chondromalacia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gamze demircioglu, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-7994
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Knee Injuries
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The rehabilitation group. (Experimental): rehabilitation group.
  Interventions: Other: The experimental group.
- The home exercise group (Active Comparator): The home exercise group
  Interventions: Other: The home exercise group

INTERVENTIONS:
Other: The experimental group. — In the experimental group, in addition to home exercises, patella mobilization, muscle strengthening exercises, range of motion exercises and home exercises will be performed 3 days a week for 3 sessions with a therapist.
  Arms: The rehabilitation group.
Other: The home exercise group — Participants in both groups will be included in a 3-week treatment programme.
  Arms: The home exercise group

SUMMARY:
Chondromalacia patella (CMP) is a common condition in patients presenting to healthcare units with anterior knee pain (1).

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is the most common type of pain in runners with a prevalence of 17%; it is limited to the anterior knee or the area behind the patella between the edges of the patella. Although PFPS and CMP are often considered to be the same disease, there is still controversy about the subject. It is caused by decreased quadriceps muscle strength, change in mechanical loading, lower limb kinematics and differentiation in muscle activation patterns during running .

ELIGIBILITY:
Inclusion criteria:

* 18-65 years of age.
* Being diagnosed with chondromalacia
* Participate in the work on a voluntary basis
* Obtaining informed consent from them

Exclusion criteria:

* Fracture, ligament or muscle tear in the lower extremity within the last 3 months.
* Having a systemic disease
* Having a serious injury in the last 3 months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
WOMAC | 3 weeks
  The Turkish version of the WOMAC scale will be used to evaluate the pain, stiffness and physical function of the individuals included in the study. The score of each section is calculated within itself and the total score varies between 0 and 100. High scores indicate an increase in pain and stiffness and impairment in physical function (12,13).
Stair climbing test | 3 weeks
  Stair ascent and descent test: The patient's ascent and descent time of the 11-step staircase with a height of 14 cm and a depth of 29 cm were recorded separately with a stopwatch.
Range of motion of the joint | 3 weeks
  Knee joint range of motion will be measured with a goniometer.
Star balance test | 3 weeks
  The test is a simple but time-consuming test in terms of its application and is used to measure dynamic postural balance (1). The test is based on the ability to reach the farthest possible distance on the supporting leg with the free foot in 8 different directions
Horizontal jump test | 3 weeks
  They jump to the farthest distance they can jump using their single and double legs and the best result obtained after at least 2 trials is recorded in cm. In this test, it should be noted that when contact with the ground after the jump, the measurement should be made at the heel level of the back foot, which is close to the starting line. Another point to be considered is that the participant should be stationary at the starting line. The participant cannot come to the line running and jump. But it is allowed to make a springing movement in front of the line

CONTACTS AND LOCATIONS:
Locations (1):
- Gamze Demircioğlu, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No